CLINICAL TRIAL: NCT02941796
Title: An Open-label, Randomized, Single-dose Crossover Study to Compare the Pharmacokinetics and Safety After Administration of HCP1105 Alone and Co-administration of HGP0918 and HGP0816 in Healthy Adult Subjects
Brief Title: Pharmacokinetics and Safety of HCP1105 and Co-administration of HGP0918, HGP0816 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROMA-106
Record Dates: First submitted 2016-10-11; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): T → R
  T : HCP1105 4cap R : HGP0918 4cap + HGP0816 4tab
  Interventions: Drug: HCP1105; Drug: HCP0918; Drug: HCP0816
- Sequence 2 (Experimental): R → T
  T : HCP1105 4cap R : HGP0918 4cap + HGP0816 4tab
  Interventions: Drug: HCP1105; Drug: HCP0918; Drug: HCP0816

INTERVENTIONS:
Drug: HCP1105
Drug: HCP0918
Drug: HCP0816

SUMMARY:
To investigate the pharmacokinetic properties and safety after administration of HCP1105 and co-administration of HGP0918, HGP0816 in healthy male volunteers

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetic properties and safety after administration of HCP1105 and co-administration of HGP0918, HGP0816 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing
* Healthy male volunteers, aged 19 to 55 years.
* The result of Body Mass Index(BMI) is not less than 18.5 kg/m2 , no more than 27.0 kg/m2

Exclusion Criteria:

* •Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system

  * Someone has a declined liver function and Liver enzyme (AST, ALT or total bilirubin) level exceeds more than one and a half times normal upper range
  * Somenone has a declined kidney function and his eGFR < 60mL/min/1.73m2

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
baseline-corrected Cmax of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
baseline-corrected AUCt of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
Cmax of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
AUCt of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)

SECONDARY OUTCOMES:
Cmax of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
AUCt of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
Tmax of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
t1/2β of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
baseline-corrected partial AUC12/24/48 of DHA total lipid & EPA total lipid | -20, -16, -12, 0(predose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72hr (Total 16)
AUC∞ of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
Tmax of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
t1/2β of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
CL/F of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)
Vdz/F of Rosuvastatin | 0(predose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72hr (Total 13)

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea